CLINICAL TRIAL: NCT01666457
Title: The Impact of Implementing an Infant Driven Feeding Program on Oral Feeding and Growth Outcomes of Medically Fragile Infants in the NICU
Brief Title: Impact of Implementing an Infant Driven Feeding Program on Oral Feeding and Growth Outcomes of Medically Fragile Infants in the Neonatal ICU (NICU)
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Susan M Horner, MS, APN/CNS, RNC-NIC, Developmental Specialist, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2009-13949 Horner
Record Dates: First submitted 2012-08-13; First posted 2012-08-16 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Oral Feeding Outcomes; Growth; Length of NICU Stay
Keywords: Supporting Oral Feeding in Fragile Infants (SOFFI); Infant Oral Feeding; Infant Growth; Preterm infant oral feeding; Preterm infant growth; Neonatal Intensive Care Unit (NICU)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-SOFFI infants: Infants discharged from the NICU prior to the implementation of the SOFFI infant driven feeding program with NICU staff.
- Post SOFFI infants: Subject infants discharged from the NICU at least 6 months after the implementation of the SOFFI infant driven feeding program and
  Interventions: Other: SOFFI

INTERVENTIONS:
Other: SOFFI — NICU nursing and multidisciplinary staff were trained to use the SOFFI infant driven feeding program. A small group of learners (20) were trained as resources via a 2-day course and the entire nursing staff received training during a 1-1.5 hour training lecture during their annual competencies.
  Other Names: Supporting Oral Feedings in Fragile Infants
  Groups: Post SOFFI infants

SUMMARY:
The specific aim of this pre-post trial is to compare data regarding oral feeding, length of stay, and growth outcomes of 100 NICU infants to these same outcomes following the implementation of a developmentally supportive, infant driven feeding program with the NICU staff, specifically the Supporting Oral Feeding in Fragile Infants (SOFFI) infant feeding program on a second sample of 100 NICU infants at Children's Memorial Hospital.

The specific research questions considered in this study are:

1. What is the impact of implementing the SOFFI on the oral feeding outcomes of medically fragile infants in the NICU at discharge and at 3 months post-term?
2. What is the impact of implementing the SOFFI on the growth outcomes of medically fragile infants in the NICU at discharge and at 3 months post-term?
3. What is the impact of implementing the SOFFI on the length of stay of medically fragile infants in the NICU?
4. What is the impact of implementing the SOFFI on the clarity and consistency of NICU staff evaluations and communications related to managing oral feedings with medically fragile infants?

ELIGIBILITY:
Inclusion Criteria:

* Infants of all gestations and diagnostic groups in this tertiary level NICU will be included in the sample

Exclusion Criteria:

* Infants with medical diagnoses known to impact sucking and swallowing
* Infants unable to manage their oral secretions
* Infants who remain hospitalized beyond 3 months adjusted age

  * Infants who expire or are transferred to another inpatient unit or hospital/facility prior to discharge from the NICU

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Convenience sample of NICU infants discharged home prior to the implementation of the SOFFI will be compared to a convenience sample of NICU infants discharged home following the implementation of the SOFFI.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Oral feeding outcomes | Up to 3 months
  Defined as percentage of ordered full feeding volume as ordered by NICU staff taken orally at NICU discharge and, if applicable, the number of days to take 100% of ordered feeding volume orally.
Oral Feeding Outcomes | Up to 5 months
  Infant oral feeding outcomes per structured parent phone interview at home.

SECONDARY OUTCOMES:
Growth outcomes | Up to 3 months
  Defined as an infant's height, weight and length percentiles on the Center for Disease Control (CDC) growth chart at NICU discharge
Growth Outcomes | Up to 5 months
  Growth outcomes per parent report during phone interview at home include current weight to be reported as percentile on CDC growth chart.

OTHER OUTCOMES:
Length of Stay | Up to 3 months
  Length of stay in days in the NICU
Change in NICU staff evaluations and communications r/t infants' oral feeding pre-SOFFI to post-SOFFI | Up to 2 years
  Measured by staff surveys done prior to and at least 3 months following SOFFI training with NICU staff. Two surveys include one for Registered Nurses (RNs)and second survey for MD/Advanced Practice Nursing (APN) staff.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Horner, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois, United States